CLINICAL TRIAL: NCT04567745
Title: Clinical Validation of an Automated Retinal Image Analysis System (EyeQuant) for Computation of Vascular Biomarkers Indicating Cognitive Decline
Brief Title: Automated Retinal Image Analysis System (EyeQuant) for Computation of Vascular Biomarkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Eyenuk, Inc. (Industry); Malavika Bhaskaranand PhD (Unknown); Kaushal Solanki (Unknown)
Responsible Party: Principal Investigator, Oana M. Dumitrascu, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-007289
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Vascular Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive diagnosis (Other)
  Interventions: Diagnostic Test: Retinal fundus photography

INTERVENTIONS:
Diagnostic Test: Retinal fundus photography — Fundus photographs

SUMMARY:
This study aims to provide clinical validation of EyeQuant, a fully automated retinal image analysis system for computation of vascular biomarkers indicative of cognitive disorders, using retinal fundus photographs collected from patients with mild cognitive impairment, Alzheimer's disease, and vascular dementia.

ELIGIBILITY:
Inclusion Criteria:

- Patients older than 18 years and diagnosed with mild cognitive impairment (MCI), Alzheimer's disease (AD), or vascular cognitive impairment and/or dementia (VaD).

Exclusion Criteria:

* Children and subjects with other diagnoses than those mentioned in the inclusion criteria.
* Patients without the means to visit the clinic on the assigned dates.
* Patients who are pregnant or are expecting to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
retinopathy features identification | 12 months
  The retinal vascular parameters computed using EyeQuant will be compared against the current gold-standard, based on expert annotations

CONTACTS AND LOCATIONS:
Overall Officials: Oana Dumitrascu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials